CLINICAL TRIAL: NCT06049927
Title: An Randomized, Double-blind, Controlled Phase III Clinical Trial to Evaluate the Safety and Immunogenicity of Quadrivalent Influenza Vaccine in Healthy Subjects Aged 6 to 35months
Brief Title: A Phase III Clinical Trial of Quadrivalent Influenza Vaccine in Healthy Subjects Aged 6 to 35 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-QINF-3005
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Seasonal Influenza
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group of quadrivalent influenza vaccine(0.25ml) (Experimental): 1100 subjects phase III will receive two doses of quadrivalent influenza vaccine(0.25ml) according to the immunization schedule of day 0,28
  Interventions: Biological: Quadrivalent influenza vaccine(0.25ml)
- Experimental Group of quadrivalent influenza vaccine(0.5ml) (Experimental): 1100 subjects phase III will receive two doses of quadrivalent influenza vaccine(0.5ml) according to the immunization schedule of day 0,28
  Interventions: Biological: Quadrivalent influenza vaccine(0.5ml)
- Control Group of trivalent influenza vaccine(BV) (Active Comparator): 550 subjects phase III will receive two doses of trivalent influenza vaccine(BV) according to the immunization schedule of day 0,28.
  Interventions: Biological: Trivalent influenza vaccine(BV)
- Control Group of trivalent influenza vaccine(BY) (Active Comparator): 550 subjects phase III will receive two doses of trivalent influenza vaccine(BY) according to the immunization schedule of day 0,28.
  Interventions: Biological: Trivalent influenza vaccine(BY)

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine(0.25ml) — 7.5 ug hemagglutinin (HA) of each of the four influenza strains in 0.25 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per njection.The routine of administration is Intramuscular injection into deltoid region.And the immunization schedule is two doses on day 0, 28.
  Arms: Experimental Group of quadrivalent influenza vaccine(0.25ml)
Biological: Quadrivalent influenza vaccine(0.5ml) — 15 ug hemagglutinin (HA) of each of the four influenza strains in 0.5 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per njection.The routine of administration is Intramuscular injection into deltoid region.And the immunization schedule is two doses on day 0, 28.
  Arms: Experimental Group of quadrivalent influenza vaccine(0.5ml)
Biological: Trivalent influenza vaccine(BV) — 7.5μg inactivated influenza antigen (H1N1, H3N2, Victoria) of each of the trivalent influenza vaccine in 0.25 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.The routine of administration is Intramuscular injection into deltoid region. And the immunization schedule is two doses on day 0, 28.
  Arms: Control Group of trivalent influenza vaccine(BV)
Biological: Trivalent influenza vaccine(BY) — 7.5μg inactivated influenza antigen (H1N1, H3N2, and Yamagata) of each of the trivalent influenza vaccine in 0.25 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.The routine of administration is Intramuscular injection into deltoid region.And the immunization schedule is two doses vaccine on day 0, 28.
  Arms: Control Group of trivalent influenza vaccine(BY)

SUMMARY:
A phase III clinical trial of the study of quadrivalent influenza vaccine developed by Sinovac Biotech will be conducted in Chinese children aged 6 to 35 months. The trial is an randomized, double-blind and active controlled study. The objective of this study is to evaluate the Immunogenicity and safety of the vaccine.

DETAILED DESCRIPTION:
A phase III clinical trial of the study of quadrivalent influenza vaccine developed by Sinovac Biotech will be conducted in Chinese children aged 6 to 35 months. The trial is an randomized, double-blind and active controlled study. The objective of this study is to evaluate the safety and immunogenicity of quadrivalent influenza vaccine(0.25ml and 0.5ml) manufactured by Sinovac Biotech Co., Ltd in healthy infants aged from 6 to 35 months. A total of 3300 subjects will be enrolled. The subjects will be randomly assigned to 4 groups in a 2:2:1:1 ratio and subjects will receive two doses of quadrivalent influenza vaccine(0.25ml or 0.5ml) or trivalent influenza vaccine(BV or BY), respectively, according to the immunization schedule of day 0,28 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 6-35 months;
* Proven vaccination certificate and birth certificate;
* The subjects' guardians can understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* Received any circulating seasonal influenza vaccine prior to enrollment or had an influenza vaccine schedule during the study;
* Suffering from seasonal influenza in the past 6 moths;
* Axillary temperature >37.0°C;
* History of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, angioedema and asthma;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Severe chronic diseases(Such as down syndrome, diabetes, sickle cell anaemia or neurological disorders);
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Autoimmune disease (such as systemic lupus erythematosus) or immunodeficiency / immunosuppression (such as HIV, after organ transplantation)
* Thyroid disease or history of thyroidectomy, asplenia,functional asplenia, asplenia or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Continuous use of corticosteroids or other immunosuppressive agents for ≥ 14 days within the past 6 months (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) and cytotoxic therapy in the past 6 months;
* Acute diseases or acute exacerbation of chronic diseases in the past 3 days;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Participated in other clinical trials before enrollment and in the follow-up period, or plans to participate in other clinical trials during the clinical trial;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3300 (Actual)
Dates: Start 2023-09-16 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates of HI antibody | 28 days after full schedule immunization
  Anti-influenza antibodies were measured using HAI assay for 4 strains: H1N1, H3N2, B Victoria and B Yamagata. Seroconversion was defined as pre-vaccination titer <1：10 and post-vaccination titer ≥1:40, and Significant increase was defined as pre-vaccination titer≥1:40 and ≥ 4-fold increase of post-vaccination titer.
Geometric Mean Titers (GMTs) of HI antibody | 28 days after full schedule immunization
  Anti-influenza antibody levels were measured using hemagglutination inhibition (HAI) assay for 4 strains: H1N1, H3N2, B Victoria, B Yamagata.
Number of Participants With Seroprotection to Influenza Vaccine Antigens | 28 days after full schedule immunization
  Anti-influenza antibodies were measured using HAI assay for 4 strains: H1N1, H3N2, B Victoria and B Yamagata. Seroprotection was defined as an antibody titer ≥1:40 at pre-vaccination and at post-final vaccination.

SECONDARY OUTCOMES:
GMIs of HI antibody | 28 days after full schedule immunization
  Anti-influenza antibody were measured using hemagglutination inhibition (HAI) assay for 4 strains: H1N1, H3N2, B Victoria, B Yamagata. GMI is the increase fold of GMT post vaccination compared with pre vaccination
Incidence of adverse reactions | 0-30 days after each dose
  Incidence of adverse reaction 0-30 days after each dose
Incidence of adverse reactions | 0-7 days after each dose
  Incidence of adverse reaction 0-7 days after each dose
Incidence of Serious adverse events | Since the beginning of vaccination until 6 months after the last dose
  Incidence of serious adverse events from beginning of vaccination until 6 months after the last dose
Incidence of AESI | since the beginning of vaccination until 6 months after the last dose
  Incidence of AESI since the beginning of vaccination until 6 months after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Lei Wang, Principal Investigator — Hubei Provincial Center for Disease Prevention and Control; Jihai Tang, Principal Investigator — Anhui Provincial Center for Disease Prevention and Control
Locations (5):
- China (5):
  - Huoqiu County Center for Disease Control and Prevention, Lu'an, Anhui
  - Zhushan County Center for Diseases Control and Prevention, Shiyan, Hubei
  - Nanzhang County Center for Disease Prevention and Control, Xiangyang, Hubei
  - Laohekou Center for Disease Control and Prevention, Xiangyang, Hubei
  - Zigui County Center for Disease Control and Prevention, Yichang, Hubei

REFERENCES:
- [Derived] Wang L, Li L, Yang W, Pang X, Li D, Zhu T, Wang S, Li T, Tian Y, Jiang Z, Li J, Yang X, Zhao C, Tang J, Tong Y. Immunogenicity and safety of inactivated quadrivalent influenza vaccines in children aged 6-35 months: A multi-center, randomized, double-blind, active-controlled clinical trial. Vaccine. 2026 Jan 25;71:128113. doi: 10.1016/j.vaccine.2025.128113. Epub 2025 Dec 13. PMID 41391373

DOCUMENTS (2):
  • Study Protocol (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT06049927/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT06049927/SAP_001.pdf